CLINICAL TRIAL: NCT03738930
Title: Effectiveness of Artificial Intelligent Based mHealth System(Chronic Disease Management System) to Reduce ACS Patients Bleeding Events After PCI: Parallel Randomized Controlled Trial
Brief Title: Effectiveness of Artificial Intelligent Based mHealth System to Reduce ACS Patients Bleeding Events After PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AI-mHealth-pilot
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Bleeding
Keywords: Acute Coronary Syndrome; Percutaneous coronary intervention; Bleeding
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal follow-up group (No Intervention): normal follow-up in ACS patients after PCI
- AI based mHealth system follow-up group (Experimental): AI based mHealth system follow-up in ACS patients after PCI. ACS patients in this group will receive message to take more notice to bleeding events.
  Interventions: Behavioral: AI based mHealth system

INTERVENTIONS:
Behavioral: AI based mHealth system — AI based mHealth system is used to deliver self-management contral message and health education message to make patients take notice of bleeding events after PCI.
  Arms: AI based mHealth system follow-up group

SUMMARY:
The present study was designed to observe the effectiveness of artificial intelligent based mHealth system(Chronic disease management system) to reduce bleeding events in ACS patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

age≥18 years, male or female; confirmed acute coronary syndrome patients; undergo percutaneous coronary intervention (PCI) treatment; good command of smart phones agree to participate in this clinical study and sign a written consent form.

Exclusion Criteria:

ACS admission deemed secondary to other cause such as traffic accidents, trauma, severe upper gastrointestinal bleeding, surgery, or procedure; patients who are not intend to attend 1 year of follow-up study or investigators find that patients are not able to comply with the study's requirements; pregnant women or lactating women; investigators consider patients who were not suitable for participation with other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2018-11-10 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of major bleeding during each visit between normal group and smartphone based group | 3 months
  Bleeding definition：According to the bleeding Academic Research Congress (BARC) standard

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Master, Principal Investigator — The General Hospital of PLA
Locations (1):
- The General Hospital of PLA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided